CLINICAL TRIAL: NCT04083209
Title: Effect of Preoperative Counseling on Postoperative Opioid Use Following Knee Arthroscopy. A Randomized Controlled Trial.
Brief Title: Effect of Preoperative Counseling on Postoperative Opioid Use Following Knee Arthroscopy.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Indiana University (Other)
Responsible Party: Principal Investigator, Robert Gerald Klitzman, Principal Investigator, Assistant Clinical Professor, Indiana University
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: 1001
Record Dates: First submitted 2019-09-06; First posted 2019-09-10 (Actual); Last update posted 2021-05-14 (Actual); Status verified 2021-05

CONDITIONS: Opioid Use; Opioid-use Disorder
MeSH Terms: conditions — Opioid-Related Disorders

STUDY DESIGN:
Intervention Model Description: Patients will be randomized into a treatment and control group.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Counseling group (Experimental): Patients randomized into the "counseling group" will be given a 1-2 minute presentation over the risks of opioid pain medications during their preoperative visit.
  Interventions: Behavioral: Opioid counseling
- Control group (No Intervention): The control group will undergo the standard preoperative evaluation by the senior author without any additional formal opioid counseling.

INTERVENTIONS:
Behavioral: Opioid counseling — The formal opioid counseling will involve reading the recommendations for postoperative opioid use established by the Pennsylvania Orthopedic Society.
  Arms: Counseling group

SUMMARY:
Our study looks to evaluate the effect of brief preoperative counseling on opioid use following knee arthroscopy. We aim to quantify the effect we have as providers in changing patient behavior postoperatively in terms of the type and amount of pain medication that is utilized.

DETAILED DESCRIPTION:
Amid a national opioid epidemic, providers are looking for ways to minimize the utilization of narcotic and addictive pain medications while adequately treating acute and postoperative pain, all the while maintaining patient satisfaction. Much effort has been dedicated to studying non-narcotic alternative medications such as acetaminophen, NSAIDs, toradol, ketamine, ect., as well as multimodal strategies such as periaxial and perineural blockades. Little attention, however, has been given to the role we play as providers to help minimize the use of these addictive medications and the potential effect we have on changing patient behaviors. Alter et al1 published in the Journal of Hand Surgery their success of minimizing opioid use by simple preoperative counseling of patients undergoing carpal tunnel release surgery. They provided brief educational materials about the opioid epidemic and risks of these medications, as well as encouraging patients to utilize non-narcotic alternatives to control pain postoperatively. They saw a decrease in the amount of opioids used with no difference in pain scores in the group receiving this preoperative counseling.

There are roughly 750,000 knee scopes performed each year in the United States. The incidence of chronic opioid use stemming from a short course of narcotics after elective knee arthroscopy has been shown to be up to 30%.2-4 The high volume of these procedures presents a unique opportunity to study trends in opioid use and pain control in the postoperative period in a prospective fashion.

Study Design

Patients scheduled to undergo knee arthroscopy by a single surgeon will be randomized into preoperative counseling or no counseling by simple randomization methods (computer generated "coin flip"). Those in the counseling group will receive a two minute talk during their preoperative appointment covering the risks of opioid medications, current public health situation regarding opioids, and alternative methods for pain control. They will also receive a one page document summarizing the Pennsylvania Orthopedic Society recommendations regarding opioid use that was used in previous research1. All patients will be prescribed the same pain medication and quantity (hydrocodone-acetaminophen 5-325 mg, 40 pills, 0 refills). Postoperatively, patients will be contacted via telephone on postoperative day three, asking what medication and how many pills they are taking daily for pain, as well as rating their daily pain level on a scale from 0-10. At their first postoperative follow-up appointment, they will again be asked about the quantity of pain medications used and pain level. After the first postoperative phone call, all data collection will be obtained at their regularly scheduled postoperative office visits, which occur at two and four weeks postoperatively. During all postoperative data collection time points we will also inquire and note all pain control measures, including ice, heat, compression, elevation, or other medications not commonly thought of as "pain medications". Data collection from each patient will be concluded at their one month postoperative visit.

ELIGIBILITY:
Inclusion Criteria:

* Patients aged 18-60, undergoing knee arthroscopic meniscectomy surgery

Exclusion Criteria:

* Non-english speaking, prisoners, those who cannot provide consent on their own, previous history of chronic opioid use, prior history of surgery on the ipsilateral knee, and those undergoing additional surgical procedures on the same knee at the time of the surgery

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 43 (Actual)
Dates: Start 2019-10-15 (Actual); Primary Completion 2020-06-26 (Actual); Study Completion 2020-06-26 (Actual)

PRIMARY OUTCOMES:
Quantity of opioid pain medication used | 2 weeks
  Patients will be tracked for the amount of opioid pain medication that is used during their postoperative course using a pill log.

SECONDARY OUTCOMES:
VAS pain scores | 2 weeks
  Patients will also be surveyed on their pain level postoperatively using the VAS pain scale. The scale is from 0-10 with 10 being the highest amount of pain. 0 representing no pain.

CONTACTS AND LOCATIONS:
Overall Officials: Mitch Beckert, MD, Principal Investigator — Indiana University School of Medicine
Locations (1):
- IU Methodist Hospital, Indianapolis, Indiana, United States

IPD SHARING:
Plan to Share IPD: Undecided
We plan to share all data collected from the study including non-identifiable patient demographics, pain scores, opioid medication utilization, complications, and study design.

REFERENCES:
- [Result] Tepolt FA, Bido J, Burgess S, Micheli LJ, Kocher MS. Opioid Overprescription After Knee Arthroscopy and Related Surgery in Adolescents and Young Adults. Arthroscopy. 2018 Dec;34(12):3236-3243. doi: 10.1016/j.arthro.2018.07.021. Epub 2018 Nov 2. PMID 30396797
- [Result] Rozet I, Nishio I, Robbertze R, Rotter D, Chansky H, Hernandez AV. Prolonged opioid use after knee arthroscopy in military veterans. Anesth Analg. 2014 Aug;119(2):454-459. doi: 10.1213/ANE.0000000000000292. PMID 24977636
- [Result] Alter TH, Ilyas AM. A Prospective Randomized Study Analyzing Preoperative Opioid Counseling in Pain Management After Carpal Tunnel Release Surgery. J Hand Surg Am. 2017 Oct;42(10):810-815. doi: 10.1016/j.jhsa.2017.07.003. Epub 2017 Sep 8. PMID 28890331